CLINICAL TRIAL: NCT04953793
Title: High School SUCCESS: Vocational Soft Skills Program for Transition-Age ASD Youth
Acronym: TAY SUCCESS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Rady Children's Hospital, San Diego (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R34MH111491 (NIH)
Record Dates: First submitted 2021-06-11; First posted 2021-07-08 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-06

CONDITIONS: Autism Spectrum Disorder
Keywords: executive functioning; social cognitions; social communication; transition age youth
MeSH Terms: conditions — Autism Spectrum Disorder; Communication

STUDY DESIGN:
Intervention Model Description: A small feasibility randomized clinical trial with randomization occurring at school site level. Two sites randomized to intervention and two sites randomized to control conditions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TAY SUCCESS intervention (Experimental): This intervention group received the TAY SUCCESS intervention over the course of 1 school year approximately 30 sessions.
  Interventions: Behavioral: TAY SUCCESS
- Usual Care (Active Comparator): This usual care group received typical High school or transition program curriculum over the course of 1 school year.
  Interventions: Other: Usual Care

INTERVENTIONS:
Behavioral: TAY SUCCESS — TAY SUCCESS stands for transition age youth supported, comprehensive cognitive enhancement and social skills. The cognitive-behavioral intervention teaches a number of strategies for executive functioning, social cognitive functioning and social communication.
  Arms: TAY SUCCESS intervention
Other: Usual Care — Usual care involved the typical vocational supportive education program delivered in the educational setting
  Arms: Usual Care

SUMMARY:
By utilizing community-based participatory research methods, this research was conducted in collaboration with the community through our partnership of researchers, educators, providers and consumers (Active Collaborative Hub for Individuals with ASD to Enhance Vocation and Education- ACHIEVE) to adapt a vocational soft skills program, Supported, Comprehensive Cognitive Enhancement & Social Skills (SUCCESS), for Transition Age Youth (TAY). The first step (years 1-2) involved adapting the intervention for autistic TAY by including feedback from multiple stakeholders and developing a curriculum to be implemented in both High Schools and Transition programs for the specific needs of autistic TAY and alpha piloting it. It involved understanding further the educational context for TAY students and current services available to prepare students for secondary outcomes of employment and/or college through a county wide survey. Step 2 (years 2-3) included pilot testing the feasibility, acceptability, implementation procedures and initial youth outcomes of the TAY SUCCESS intervention and further refining the curriculum and protocols. Findings demonstrated improvements in executive functioning and social functioning targets as well as distal outcomes of self-efficacy, mental health, educational and work behaviors and attitudes. The study results were disseminated through the ACHIEVE group as well as at conferences, website and publication.

DETAILED DESCRIPTION:
Aim: With our ACHIEVE partners , develop the High School Supported, Comprehensive Cognitive Enhancement and Social Skills (SUCCESS) program to fit the needs of transition-age youth with ASD within the community educational system.

1. Standardize the TAY SUCCESS program by developing a facilitator manual, student workbook and corresponding support person materials.
2. Develop a training protocol that can be individualized and implemented within the HS educational system to provide initial training and ongoing coaching for educators to reach and sustain intervention fidelity.

Aim: Conduct a pilot study to examine the feasibility, acceptability, and implementation procedures (recruitment, randomization, retention & training strategies) of TAY SUCCESS and to obtain estimates of effects to support a future large-scale effectiveness trial.

1. Examine intervention feasibility, acceptability, satisfaction, and sustainability.
2. Examine preliminary outcomes (executive functioning and social functioning)

ELIGIBILITY:
Inclusion Criteria:

* autism spectrum disorder
* 15-22 yrs
* communicative English language
* enrolled in participating high school or transition program

Exclusion Criteria:

* intellectual disability
* Other significant mental health

Ages: 15 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 42 (Actual)
Dates: Start 2017-11-06 (Actual); Primary Completion 2020-01-20 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Behavior Rating Inventory of Executive Function (BRIEF-2/BRIEF-A) | baseline to 6 month post
  Self and Parent report of executive functioning skills. Higher scores indicate more executive functioning problems
Delis Kaplan Executive Function Scale (DKEFS) | baseline to 6 month post
  performance based measure of executive functioning skills. Higher scores indicate more executive functioning abilities
Social Responsiveness Scale 2 (SRS-2) | baseline to 6 month post
  parent report social functioning scale. Higher scores indicate more social functioning problems

CONTACTS AND LOCATIONS:
Locations (1):
- Rady Children's Hospital San Diego, San Diego, California, United States

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-15): https://cdn.clinicaltrials.gov/large-docs/93/NCT04953793/Prot_SAP_000.pdf